CLINICAL TRIAL: NCT03136068
Title: Intrafetal Digoxin as an Adjuvant for Dilation and Evacuation at 20 to 24 Weeks' Gestation: a Placebo-controlled, Double-blinded Randomized Controlled Trial
Brief Title: Intrafetal Digoxin as an Adjuvant for Dilation and Evacuation at 20 to 24 Weeks' Gestation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: FPA Women's Health (Unknown); Society of Family Planning (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jennifer Kerns, MD, MS, MPH, Assistant Professor department of Obstetrics, Gynecology and Reproductive Sciences, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Digoxin RCT
Record Dates: First submitted 2017-02-06; First posted 2017-05-02 (Actual); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Abortion
MeSH Terms: interventions — Digoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Digoxin (Experimental): Subjects assigned to the intervention arm will receive a 1 mg intrafetal digoxin injection under ultrasound guidance
  Interventions: Drug: Digoxin
- Placebo (Placebo Comparator): Subjects assigned to the control arm will receive an ultrasound-guided intrafetal saline injection of the equivalent volume
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Digoxin — Trans-abdominal injection
  Arms: Digoxin
Drug: Placebo — Trans-abdominal injection
  Arms: Placebo

SUMMARY:
This is a research study to measure the effect of digoxin injection on Dilation and Evacuation (D&E) procedure duration. Digoxin is the most commonly used feticidal agent among family planning subspecialists, and is commonly used for a variety of reasons including provider preference, patient preference, and concerns over legal status of later D&E procedures. There have been several studies on digoxin administration, adverse effects, and impact on the D&E procedure, but doctors want to clarify how digoxin effects D&E procedure time, if at all.

ELIGIBILITY:
Inclusion Criteria:

* 20 weeks 0 days-24 weeks 0 days gestation
* English or Spanish speaking
* 18 years or older

Exclusion Criteria:

* Under 18
* Contraindications to digoxin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - FPA Women's Health, Long Beach, California
  - SFGH Women's Options Center, San Francisco, California
  - Lovejoy Surgicenter, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Digoxin | Placebo
Started | 88 | 90
Completed | 86 | 89
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digoxin | Placebo | Total
Number analyzed (Participants) | 88 | 90 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (6.7) | 26.2 (5.6) | 26.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 90 | 178
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian, non-Hispanic | 26 | 30 | 56
  Hispanic | 28 | 31 | 59
  African-American, non-Hispanic | 17 | 17 | 34
  Mixed/Multi | 8 | 8 | 16
  Other | 9 | 4 | 13
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.2 (5.6) | 26.7 (5.2) | 26.9 (5.4)
Nulliparous [Count of Participants; unit: Participants] | 21 | 15 | 36
Gestational duration [Median (Inter-Quartile Range); unit: weeks] | 21.1 [21 to 22] | 21.0 [20 to 22] | 21.0 [20.4 to 21.9]

OUTCOME MEASURES:

1. Primary Outcome: Procedure Duration
Description: First instrument into uterus until procedure complete
Time Frame: Beginning to end of procedure (between 5 minutes and 1 hour)
Population: Duration of procedure time from speculum insertion to procedure completion
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Digoxin | Placebo
Number analyzed (Participants) | 86 | 89
minutes | 6.8 (4.8) | 7.2 (6.9)

2. Secondary Outcome: Total Procedure Duration
Description: Time from speculum placed until all instruments removed from vagina (including speculum and fingers) and done with everything
Time Frame: done on Day 2 during the procedure
Population: duration of procedure for each participant from insertion of speculum to total procedure completion, including any post-procedure activities prior to being taken to recovery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Digoxin | Placebo
Number analyzed (Participants) | 86 | 89
minutes | 9.7 (9.3) | 8.3 (7.9)

3. Secondary Outcome: Measured Blood Loss
Description: measured blood loss, in mL, during the procedure, measured by weighing the absorbent materials used and subtracting out their weight without blood
Time Frame: Day 2, during the procedure
Population: measured blood loss was only completed at the Zuckerberg San Francisco General Hospital location, which is why the total is 61 rather than 175 for this outcome
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Digoxin | Placebo
Number analyzed (Participants) | 33 | 28
mL | 417 [305 to 527] | 363 [279 to 522]

4. Secondary Outcome: Number of Patients With Reported Fetal Death Prior to Procedure
Description: number of patients who had fetal death measured by ultrasound
Time Frame: Day 2, before procedure
Population: number of patients who had reported fetal death on day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Digoxin | Placebo
Number analyzed (Participants) | 86 | 89
Participants | 68 | 6

5. Secondary Outcome: Complications
Description: hemorrhage, perforation, cervical laceration requiring suture repair, out-of-hospital delivery, infection, inability to complete injection, other complications of the injection itself, and patient symptoms such as nausea and vomiting
Time Frame: Day 2
Population: any complication reported by patient; may have reported more than one complication
Measure: Count of Participants; unit: Participants
Arm/Group | Digoxin | Placebo
Number analyzed (Participants) | 89 | 86
Participants | 8 | 4

ADVERSE EVENTS:
Time Frame: two days, day one and day two
Description: does not differ from clinicaltrials.gov
Arm/Group | Digoxin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/86 | 1/89
Other Adverse Events (participants affected / at risk) | 7/86 | 3/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin (N=86) | Placebo (N=89)
blood transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Post-D&E hemorrhage, patient admitted for transfusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin (N=86) | Placebo (N=89)
pregnancy labor (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — patient went into labor prior to D&E (Dilation and evacuation), had D&C (Dilation and curettage)
severe nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
hemmorhage (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — 1 post-D&E hemorrhage (requiring vag pack and med tx) 1 intra-op hemorrhage requiring Foley and med tx
anxiety (Nervous system disorders) | 0 (0) | 1 (1) — severe anxiety/pain post D&E requiring medications
cramping (Reproductive system and breast disorders) | 1 (1) | 1 (1) — extreme cramping pain following injection severe cramping pain post D&E requiring medications
fever (General disorders) | 1 (1) | 0 (0)
mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) — MD identified uterine mass, pt transferred to hospital
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — extreme nausea/vomiting following injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT03136068/Prot_SAP_000.pdf